CLINICAL TRIAL: NCT06815432
Title: GPC-3 Chimeric Antigen Receptor T Cells FOR Recurrent GPC-3 Positive Glioblastoma
Brief Title: GPC-3 CAR T CELLS FOR Recurrent GPC-3 Positive Glioblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); Baylor St. Luke's Medical Center (Other)
Responsible Party: Principal Investigator, Ganesh Rao, MD, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-55707 GO-CART
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma Multiforme of Brain
Keywords: GPC3-positive tumors; GPC3-CAR T cells; Glioblastoma; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 15.GPC3-CAR T cells (Experimental): GPC3-CAR and IL15 will be administered to patients with GPC3-positive glioblastoma.
  Interventions: Genetic: 15.GPC3-CAR T cells

INTERVENTIONS:
Genetic: 15.GPC3-CAR T cells — Four different dosing schedules will be evaluated. The following dose levels will be evaluated:
  DL1: 5x10^6 DL2: 1x10^7 DL3: 5x10^7 DL4: 1x10^8

SUMMARY:
The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells.

Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T-cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat participants with cancers. They have shown promise, but have not been strong enough to cure most participants.

The study team has found from previous research that we can put a new gene (a tiny part of what makes-up DNA and carries the participants traits) into T cells that will make them recognize cancer cells and kill them. In the lab, the study team has made several genes called a chimeric antigen receptor (CAR), from an antibody called GC33. The antibody GC33 recognizes a protein found on the participants brain tumor. This CAR is called GPC3-CAR. To make this CAR more effective, the study has also added a gene that includes IL15. IL15 is a protein that helps CAR T cells grow better and stay in the blood longer so that they may kill tumors better. The mixture of GPC3-CAR and IL15 killed tumor cells better in the laboratory when compared with CAR T cells that did not have IL15. This study will test T cells with the IL15 GPC3-CAR (GO-CART T cells) in participants with GPC3-positive brain tumors.

T cells made to carry a gene called iCasp9 can be killed when they encounter a specific drug called AP1903. The study team will insert the iCasp9 and IL15 together into the T cells using a virus that has been made for this study. The drug (AP1903) is an experimental drug that has been tested in humans with no bad side-effects. The study team will use this drug to kill the T cells if necessary due to side effects.

This study will test T cells genetically engineered with a GPC3-CAR and IL15 (GO-CART T cells) in participants with GPC3-positive brain tumors.

The GO-CART T cells are an investigational product not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
The study team will collect up to 180 mL (approximately 12 tablespoons) of participants blood. This will be used to grow T cells. The study team grows the T cells and uses a retrovirus (a special virus that can insert the GPC3 CAR and IL15 genes into the T cells) to genetically engineer them. After the CAR and IL15 genes were put into the T cells, the study team ensures that they could kill GPC3 positive solid tumor cells in the laboratory.

WHAT THE TREATMENT WILL BE LIKE:

After making these cells, they were frozen. If the participant agrees to participate in this study, at the time they are scheduled to be treated, the cells will then be thawed and administered in the participants tumor area, called an intracavitary administration, during the participants already scheduled surgical resection. The participant will only get one dose of GO-CART T cells. The participant may be pretreated with Tylenol (acetaminophen) and Benadryl (diphenhydramine). Tylenol and Benadryl are given to prevent a possible allergic reaction to the T cell administration.

In addition to the GO-CART T cell treatment, during surgery the surgeon will place a small device called an Ommaya reservoir. This device consists of a small tube approximately 3 millimeters in diameter whose tip will sit in the normal fluid filled spaces in the participants brain (called the ventricles). The other end of the tube will be attached to a small reservoir that will sit underneath the participants scalp. Ommaya reservoirs are commonly placed in cancer participants to treat participants with cancer cells in the cerebrospinal fluid and pose a low risk of complications. The purpose of this reservoir is to help reduce the pressure in the participants brain should they experience this from the treatment which is an unlikely but reported side effect . The reservoir will also be used to monitor the participants response to the study treatment rather than to administer treatment.

This is a dose escalation study, which means that the study team does not know the highest dose of GO-CART T cells that is safe. To find out, the cells will be given to at least 3 participants at a lower dose. If that is safe, the study team will raise the dose level that is given to the next group of participants. The dose a participant received will get will depend on how many participants get the agent before the participant and how they react. The investigator will tell the participant this information. Since the treatment is experimental, what is likely to happen at any dose is not known.

All the treatments will be given by the Center for Cell and Gene Therapy at Baylor St. Luke's Medical Center.

Medical tests before treatment:

Before being treated, the participant will receive a series of standard medical tests:

* Physical exam and history
* Blood tests to measure blood cells, kidney and liver function.
* Pregnancy test (if the participant is a female who can get pregnant)
* If the participant is infected with the hepatitis B virus (HBV) the study team will do a test to measure the levels of the virus
* Measurements of the participants tumor by scans (either CT or MRI). Side effects are rare and include risk of developing an unrelated cancer due to radiation exposure from the machine, but this is unlikely.

Medical tests during and after treatment:

The participant will receive standard medical tests when they are getting the infusions and after:

* Physical exams and History
* Blood tests to measure blood cells, kidney and liver function.
* If the participant is infected with the hepatitis B virus (HBV) the study team will repeat the test and monitor the levels of the virus
* Cerebral spinal fluid collections to monitor for any side effects during the course of the treatment
* Measurements of the participants tumor by scans (1 week, and 4 - 6 weeks after the treatment)

FOLLOW-UP STUDIES:

The study team will follow the participant during and after the injections. To learn more about the way the T cells are working in the participants body, up to 60 mL (up to 12 teaspoons, no more than 3mL/kg/day) of blood will be taken before the chemotherapy, before the T-cell infusion, 1 to 4 hours after the infusion, 3 to 4 days after the infusion (this time point is optional) at 1 week, 2 weeks, 3 weeks, 4 weeks and 8 weeks after the injection, every 3 months for 1 year, every 6 months for 4 years and then every year for the next 10 years. Total participation time for this study will be 15 years.

During the time points listed above, if the T cells are found in the participants blood at a certain amount an extra 5mL of blood may need to be collected for additional testing.

The study team will use this blood to look for the frequency and activity of the cells that have been given ; that is, to learn more about the way the T cells are working and how long they last in the body. The study team will also use this blood to see if there are any long-term side effects of putting the new gene (chimeric antigen receptor, CAR) into the cells. In addition to the blood draws, because the participant has received cells that have had a new gene put in them, they will need to have long term follow up for 15 years to see if there are any long-term side effects of the gene transfer.

Once a year, the participant will be asked to have their blood drawn and answer questions about their general health and medical condition. The study team may ask the participant to report any recent hospitalizations, new medications, or the development of conditions or illness that were not present during enrollment in the study and may request that physical exams and/or laboratory tests be performed if necessary.

If the participants tumor requires further surgery after the study treatment, for clinical reasons the study team will request permission to obtain excess sample to learn more about the effects of the treatment on the participants disease.

In the event of death, the study team will request permission to perform an autopsy to learn more about the effects of the treatment on the participants disease and if there were any side effects from the cells with the new gene.

In addition, the study team will ask for the participants permission to use tumor biopsy for research purposes only. Associated risk with the biopsy will be discussed with the participant in detail in a procedure specific consent form. The study team will test the sample to see if the GO-CART T cells can be found in the tumor and what effect they had on the tumor cells.

If the participant develops a second abnormal cancer growth, significant blood or nervous system disorder during the trial, the study team will request that a biopsy sample of the tissue will be tested.

The remaining blood and/or tissue samples that are not needed directly for the participant could be used to help researchers learn about this disease and/or immune therapy. These specimens and information about the participants circumstances may be shared with other cancer researchers. Although there will be a record identifying under what circumstances these specimens were obtained, under all circumstances the participants identity will be kept confidential. There is a small risk for the loss of confidentiality. However, study personnel will make every effort to minimize this risk. Samples will be kept at Baylor College of Medicine until they are exhausted.

ELIGIBILITY:
Procurement Inclusion Criteria:

* Diagnosis of GPC3-positive recurrent glioblastoma with previous resection planned for repeat resection.
* Age ≥18 years
* Karnofsky score ≥60%
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent
* GPC3 expression (as determined by immunohistochemistry) with an extent score of ≥ Grade 2 (>25% positive tumor cells) and an intensity score of ≥ 2 (scale 0-4).

Procurement Exclusion Criteria:

* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies).
* History of organ transplantation
* Known HIV positivity
* Active bacterial, fungal or viral infection (except Hepatitis B or Hepatitis C virus infections).
* Exhibits other risk factors of which administration of investigational agent is deemed not in the patient's best interest, in the opinion of the investigator

Treatment Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of recurrent glioblastoma with previous resection
* Karnofsky score ≥ 60%-
* Stable neurologic exam for 7 days prior to enrollment
* Stable or decreasing dose of steroids over past 7 days prior to surgery and administration of therapy (max allowable dose is 0.1mg/kg dexamethasone or equivalent per day)
* Adequate organ function:
* Creatinine clearance as estimated by Cockcroft Gault or Schwartz ≥ 60 ml/min
* total bilirubin < 3 times ULN for age
* INR ≤1.7
* absolute neutrophil count > 500/μl
* platelet count > 100,000/μl (can be transfused but must be achieved prior to enrollment)
* Hgb ≥ 7.0 g/dl (can be transfused)
* Pulse oximetry >90% on room air
* Recovered from acute toxic effects of all prior chemotherapy and investigational agents before entering this study
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 3 months after the T-cell infusion.
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

Treatment Exclusion Criteria:

* Pregnancy or lactation
* Uncontrolled infection
* Known HIV positivity
* Active bacterial, fungal or viral infection
* History of organ transplantation
* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2029-12-05 (Estimated); Study Completion 2044-12-03 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | 4 weeks
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the 15.GPC3-CAR T cells. Specifically those which are Grade 5; hematologic dose-limiting toxicity is any Grade 4 non-hematologic toxicity that fails to return to Grade 2 within 72 hours; Grade 4 allergic reaction to CAR T cell administration; Grade 4 \reactions due to CRS and neurotoxicity are rarely seen with the use of CAR-based immunotherapy. Grade 3 cytokine release syndrome (CRS) infusion reactions and neurologic toxicity will only be reported to the FDA if they fail to return to Grade 1 within 72 hours. Grade 4 CRS and neurologic toxicities will be reported to the FDA in an expedited fashion.

SECONDARY OUTCOMES:
Response Rate | 4 weeks
  Response rates will be estimated as the percent of patients whose best response is either complete response or partial by combining the data from lesions recorded via imaging for each patient pre- and post-15.GPC3-CAR T-cell intracavitary administration. These data will be evaluated by iRANO criteria. A 95% confidence interval will be calculated for the response rate.
Maximum Tolerated Dose (MTD) | 4 weeks
  The maximum tolerated dose (MTD) is determined based on isotonic regression as specified in Liu and Yuan (PMID: 3162195). The dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate. If there is no DLT that determine a MTD, the maximum dose level will be declared as the MTD. In case the lowest dose level is determined to be too toxic and the elimination boundary is reached, no MTD will be defined for the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Rao, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor St. Luke's Medical Center, Houston, Texas, United States